CLINICAL TRIAL: NCT06385470
Title: Treatment of Cantonese Speakers With Childhood Apraxia of Speech
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: University of Vermont (Other); The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr Min Wong, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSEARS20231112001
Record Dates: First submitted 2024-04-22; First posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Childhood Apraxia of Speech
MeSH Terms: conditions — Apraxias

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DTTC treatment (Experimental): Four Cantonese-English bilingual children with be randomly assigned to receive either one of the two versions of DTTC (i.e., DTTC in Cantonese [DTTC-C] and DTTC in English [DTTC-E]) in the first 6-week treatment phase. Then, there will be a 2-week washout period followed by the second 6-week treatment phase with another version of DTTC.
  Interventions: Behavioral: Dynamic Temporal and Tactile Cueing treatment

INTERVENTIONS:
Behavioral: Dynamic Temporal and Tactile Cueing treatment — DTTC is a motor-based treatment designed for children with CAS who may have limited verbal output. It applies the principles of motor learning and focuses on speech movement gestures in the context of functional words and phrases.
  The participants will receive two versions of the DTTC treatment (i.e., DTTC in English [DTTC-E] and DTTC in Cantonese [DTTC-C]), where probe data will be collected before, during, between and after the treatment intervention.

SUMMARY:
The proposed study aims to investigate the efficacy of the Dynamic Temporal and Tactile Cueing treatment in Cantonese-English bilingual speakers with childhood apraxia of speech.

DETAILED DESCRIPTION:
Four CE children with CAS will be recruited and receive two versions of the DTTC treatment (i.e., DTTC in English [DTTC-E] and DTTC in Cantonese [DTTC-C]). After the initial assessment and baseline probe sessions, all the participants will be randomly assigned to receive either DTTC-E or DTTC-C in the first 6-week treatment phase. Then, the between-treatment probe sessions will be conducted during a 2-week washout period. This will be followed by the second 6-week treatment phase, which will be the other version of DTTC. Post-treatment probe sessions will be conducted one week and one month after completion of the second treatment.

Participants' speech productions will be transcribed and evaluated based on their accuracy in phonemes, stress, and tone. Growth curve analysis (Mirman, 2014) will be conducted to examine the group differences in the outcome measures across the treatment sessions.

ELIGIBILITY:
Inclusion Criteria:

* (1) 3;0 - 11;11 (years;months) years of age at treatment commencement;
* (2) speak both Cantonese and English: One caregiver one language for at least one year; speaking different languages at home versus school; and/or speak different languages at different times of day;
* (3) no concomitant developmental disorders including autism spectrum disorder;
* (4) no structural abnormalities that affect speech, such as cleft lip and/or palate;
* (5) no uncorrected vision impairment; and
* (6) no hearing loss;
* (7) CAS diagnosis confirmed by the research team based on the available diagnostic criteria in Cantonese speakers, which will be described in the next section

Exclusion Criteria:

-

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Phonemes accuracy | Change Before, Between, 1-week and 5-week post DTTC treatment
  Participants' performance is probe sessions will be transcribed and analysed by an independent research assistant who has experience with Cantonese and English disordered speech will undergo training in phonetic transcription. The training will include practicing transcription of Cantonese and English speech of preschool children on standardized articulation tests. The accuracy of phonemes and the following aspects will be judged by the research assistant.
Stress accuracy | Change Before, Between, 1-week and 5-week post DTTC treatment
  Participants' performance is probe sessions will be transcribed and analysed by an independent research assistant who has experience with Cantonese and English disordered speech will undergo training in phonetic transcription. The training will include practicing transcription of Cantonese and English speech of preschool children on standardized articulation tests. The accuracy of phonemes and the following aspects will be judged by the research assistant.
Tone accuracy | Change Before, Between, 1-week and 5-week post DTTC treatment
  Participants' performance is probe sessions will be transcribed and analysed by an independent research assistant who has experience with Cantonese and English disordered speech will undergo training in phonetic transcription. The training will include practicing transcription of Cantonese and English speech of preschool children on standardized articulation tests. The accuracy of phonemes and the following aspects will be judged by the research assistant.

CONTACTS AND LOCATIONS:
Overall Officials: Min Ney Wong, PhD, Principal Investigator — Study Principal Investigator
Locations (1):
- The Hong Kong Polytechnic University, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: No
The data sets generated and analyzed during this study are not publicly available due to study institutional review board data security requirements.